CLINICAL TRIAL: NCT00869869
Title: Restoration of Sleep in Heart Failure Patients
Brief Title: Melatonin Supplementation to Improve Sleep in Patients With Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled in this study. Funding ran out.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASMF-Scheer
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure; Sleep Disorders
Keywords: Heart Failure; Sleep Disorders; Melatonin; Antioxidants; Molecular Mechanisms of Pharmacological Action; Nervous System Diseases; Physiological Effects of Drugs; Vascular Diseases; Central Nervous System Depressants; Protective Agents; Pharmacologic Actions; Signs and Symptoms; Mental Disorders; Therapeutic Uses; Neurologic Manifestations; Cardiovascular Diseases; Central Nervous System Agents
MeSH Terms: conditions — Heart Failure; Sleep Wake Disorders; Nervous System Diseases; Vascular Diseases; Signs and Symptoms; Mental Disorders; Neurologic Manifestations; Cardiovascular Diseases | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- melatonin (Experimental): melatonin
  Interventions: Drug: melatonin
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin — 2.5 mg melatonin, by mouth, 1 per day, for 3-4 weeks
  Arms: melatonin
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether melatonin can improve sleep, quality of life and markers of heart failure in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure affects nearly 5 million individuals in the United States and constitutes a prime risk factor for morbidity and mortality. Beta-blockers are a class of drugs that form a critical part of the best treatment of heart failure, and thereby decrease the risk for these serious problems. Beta-blockers also lower the levels of melatonin, a hormone that has a sleep-promoting effect. Most patients with heart failure take beta-blockers and have poor sleep, which may be related to the beta-blockers' effect on melatonin levels. This study will evaluate the effectiveness of treatment with melatonin supplements in improving sleep in individuals with heart failure who are taking beta-blockers. In addition, the study will examine whether the melatonin supplements aid in improving quality of life and measures of heart failure.

Participants in this double-blind study will be randomly assigned to receive either melatonin supplements or placebo for the duration of the study.

The study will mainly take place at home, where participants will complete sleep diaries, measure blood pressure and wear a wrist watch that measures movement for 5-6 weeks. During that time there will be three visits to the hospital where plasma and urine samples will be collected and questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure NYHA Class 2 or 3
* Currently being treated with beta-blocker

Exclusion Criteria:

* Diagnosed with obstructive sleep apnea
* Using Fluvoxamine, Warfarin, Nifedipine, or Calcium Channel Blockers

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quantity assessed by actigraphy | measured during ambulatory phase

SECONDARY OUTCOMES:
Change in quality of life and heart failure biomarkers | measured during study visits

CONTACTS AND LOCATIONS:
Overall Officials: Frank A.J.L. Scheer, Ph.D., Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Scheer FA, Van Montfrans GA, van Someren EJ, Mairuhu G, Buijs RM. Daily nighttime melatonin reduces blood pressure in male patients with essential hypertension. Hypertension. 2004 Feb;43(2):192-7. doi: 10.1161/01.HYP.0000113293.15186.3b. Epub 2004 Jan 19. PMID 14732734
- [Background] Scheer FA, Czeisler CA. Melatonin, sleep, and circadian rhythms. Sleep Med Rev. 2005 Feb;9(1):5-9. doi: 10.1016/j.smrv.2004.11.004. No abstract available. PMID 15649734
- [Background] Scheer FA, Zeitzer JM, Ayas NT, Brown R, Czeisler CA, Shea SA. Reduced sleep efficiency in cervical spinal cord injury; association with abolished night time melatonin secretion. Spinal Cord. 2006 Feb;44(2):78-81. doi: 10.1038/sj.sc.3101784. PMID 16130027
- [Background] Scheer FA. Potential use of melatonin as adjunct antihypertensive therapy. Am J Hypertens. 2005 Dec;18(12 Pt 1):1619-20. doi: 10.1016/j.amjhyper.2005.07.013. No abstract available. PMID 16364835
- [Background] Scheer FA, Stone PH, Shea SA. Decreased sleep in heart failure: are medications to blame? Arch Intern Med. 2007 May 28;167(10):1098-9; author reply 1099-100. doi: 10.1001/archinte.167.10.1098-b. No abstract available. PMID 17533214